CLINICAL TRIAL: NCT04410445
Title: A Phase 3, Randomized, Open-label Study to Compare Adjuvant Immunotherapy of Bempegaldesleukin Combined With Nivolumab Versus Nivolumab After Complete Resection of Melanoma in Patients at High Risk for Recurrence (PIVOT-12)
Brief Title: Study to Compare Adjuvant Immunotherapy of Bempegaldesleukin Combined With Nivolumab Versus Nivolumab After Complete Resection of Melanoma in Patients at High Risk for Recurrence
Acronym: PIVOT-12
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: (Sponsor decision)
Sponsor: Nektar Therapeutics (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-214-29/CA045-022
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-03

CONDITIONS: Melanoma; Melanoma Stage III; Melanoma Stage IV; Melanoma (Skin)
Keywords: CD122-Biased Agonist; CD122-Biased Cytokine; IL-2 Receptor Agonist; NKTR-214; Bempegaldesleukin; IL-2; Immunotherapy; BEMPEG; Nivolumab; Opdivo®; NIVO; Adjuvant; Skin Cancer; Resectable Melanoma; High Risk of Recurrence Melanoma; Post Resection; Checkpoint Inhibitor
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — bempegaldesleukin; Nivolumab

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio to one of two treatment arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Combination of bempegaldesleukin (NKTR-214) + nivolumab (Experimental): Arm A: Participants will receive bempegaldesleukin (NKTR-214) IV in combination with nivolumab every 3 weeks.
  Interventions: Biological: Bempegaldesleukin; Biological: Nivolumab
- Nivolumab (Active Comparator): Arm B: Participants will receive nivolumab IV alone every 4 weeks.
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Bempegaldesleukin — Specified dose on specified days
  Other Names: NKTR-214; BMS-986321
  Arms: Combination of bempegaldesleukin (NKTR-214) + nivolumab
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo®; BMS-936558

SUMMARY:
The main purpose of this study is to compare the efficacy of bempegaldesleukin plus nivolumab versus nivolumab in patients with completely resected Stage IIIA/B/C/D, or Stage IV cutaneous melanoma who are at high risk for recurrence.

DETAILED DESCRIPTION:
The main purpose of this study is to compare the efficacy, as measured by recurrence-free survival (RFS) by blinded independent central review (BICR), of bempegaldesleukin plus nivolumab versus nivolumab in patients with completely resected Stage IIIA (lymph node [LN] metastasis > 1 mm), Stage IIIB/C/D, or Stage IV (American Joint Committee on Cancer [AJCC] 8th edition) cutaneous melanoma with no evidence of disease (NED) who are at high risk for recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age 12 years or older at the time of signing the informed consent form (age 18 years or older where local regulations, countries, and/or institutional policies do not allow for patients < 18 years of age (adolescents) to participate). In regions where adolescents are not allowed to participate in the study due to age restrictions, enrolled patients must be ≥ 18 years of age.
* Histologically confirmed Stage IIIA (LN metastasis > 1 mm), IIIB/C/D, or IV (M1a/b/c/d) cutaneous melanoma by AJCC (8th edition) at study entry that has been completely surgically resected within 12 weeks prior to randomization.
* Tumor tissue available from biopsy or resected disease must be provided to central laboratory for PD-L1 status analysis. Must have PD-L1 expression classification for stratification purposes.
* Disease-free status documented by a complete physical examination and imaging studies within 28 days prior to randomization.

Exclusion Criteria:

* History of ocular/uveal melanoma or mucosal melanoma.
* Active, known or suspected autoimmune disease. Patients with Type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Conditions requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Prior therapy for melanoma except surgery for the melanoma lesion(s) and/or adjuvant radiation therapy for central nervous system lesions.
* Prior therapy with interferon, talimogene laherparepvec (Imylgic®), interleukin-2 (IL-2) directed therapy, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T lymphocyte-associated protein 4 antibody (including ipilimumab or any other antibody or drug specifically targeting T cell co-stimulation or checkpoint pathways).
* Prior malignancy active within the previous 3 years except for locally potentially curable cancers that have been apparently cured.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 765 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (212):
- United States (62):
  - Honor Health, Scottsdale, Arizona
  - Banner MD Anderson Cancer Center, Little Rock, Arkansas
  - Kaiser Foundation Hospital, Inpatient Pharmacy, Anaheim, California
  - Kaiser Permanente, Fontana, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Hematology Oncology Medical Group of Orange County, Inc., Orange, California
  - University of California Irvine, Orange, California
  - Emad Ibrahim, MD, Inc, Redlands, California
  - Kaiser Permanente, Riverside, California
  - Southern California Permanente Medical Group, Riverside, California
  - San Francisco Oncology Associates, San Francisco, California
  - California Cancer Associates for Research and Excellence, San Marcos, California
  - Kaiser Permanente, San Marcos, California
  - Angeles Clinic and Research Institute, Santa Monica, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Rocky Mountain Cancer Centers (Littleton) - USOR, Aurora, Colorado
  - University of Colorado - Cancer Center - PPDS, Aurora, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Orlando Health Cancer Institute, Longwood, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Goshen Center For Cancer Care, Goshen, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic - PIN, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Frontier Cancer Center and Blood Institute, Billings, Montana
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Atlantic Health System, Morristown, New Jersey
  - NYU Langone Medical Center, New York, New York
  - Columbia University Medical Center - PIN, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence Cancer Institute, Franz Clinic, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Physician Group (LVPG) - Hematology Oncology, Allentown, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Jefferson University Hospital, Philadelphia, Pennsylvania
  - H Lee Moffitt Cancer Center and Research Institute, Pittsburgh, Pennsylvania
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - SCRI Tennessee Oncology Nashville, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Department of Pharmacy Investigational Drug Services, Dallas, Texas
  - Texas Oncology (Loop) - USOR, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Utah Cancer Specialists (Salt Lake City), Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Blue Ridge Cancer Care - USOR, Roanoke, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington
  - University of Wisconsin, Madison, Wisconsin
- Australia (13):
  - Royal Adelaide Hospital, Adelaide
  - Cairns Hospital, Cairns
  - Icon Cancer Care Wesley, Chermside
  - Gallipoli Medical Research Foundation, Greenslopes
  - Austin Health, Heidelberg
  - Alfred Hospital, Melbourne
  - Affinity Clinical Research, Nedlands
  - Sir Charles Gairdner Hospital, Nedlands
  - Melanoma Institute Australia, North Sydney
  - Gold Coast University Hospital, Southport
  - Tasman Oncology Research, Southport
  - Blacktown Hospital, Westmead
  - Princess Alexandra Hospital, Woolloongabba
- Austria (6):
  - Medizinische Universität Graz, Graz
  - Ordensklinikum Linz, Krankenhaus der Elisabethinen GmbH, Lienz
  - Landeskrankenhaus Feldkirch, Rankweil
  - Salzburger Landeskliniken, Salzburg
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
- Czechia (7):
  - Mou/Mmci - Ppds, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Krajska nemocnice Liberec, a.s., Liberec
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava Poruba
  - Vseobecna Fakultni Nemocnice V Praze, Prague
  - Nemocnice Na Bulovce, Prague
- France (16):
  - Centre Hospitalier Universitaire (CHU) Amiens-Picardie - Hopital Sud, Amiens
  - CHU Angers, Angers
  - Hôpital Saint-André, Bordeau
  - CHRU de Tours, Chambray-lès-Tours
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Albert Michallon La Tronche, La Tronche
  - CHRU Lille, Lille
  - Hôtel Dieu - Nantes, Nantes
  - CHU de Nice, Nice
  - Hôpital Saint Louis, Paris
  - Groupe Hospitalier Bichat Claude Bernard, Paris
  - Hospices Civils de Lyon, Pierre-Bénite
  - EDOG - Centre Eugene Marquis Centre Regional de Lutte Contre Le Cancer - PPDS, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Centre Hospitalier Universitaire de Saint Etienne, Saint-Priest-en-Jarez
  - Institut Gustave Roussy, Villejuif
- Germany (25):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Ruhr Universität Bochum, Bochum
  - Elben Klinken Stade - Buxtehude, Buxtehude
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - Universitätsklinikum Essen, Essen
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Universitatsklinikum Halle (Saale), Halle
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - University Clinic Heidelberg, Heidelberg
  - SLK Kliniken Heilbronn GmbH, Heilbronn
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - Universitatsklinikum Leipzig, Leipzig
  - Klinikum der Stadt Ludwigshafen gGmbH, Ludwigshafen
  - Universitätsklinik Magdeburg, Magdeburg
  - Klinikum Mannheim Universitätsklinikum gGmbH, Mannheim
  - Universitatsklinikum Munster, Münster
  - Fachklinik Hornheide, Münster
  - University Clinic Regensburg, Regensburg
  - Helios Klinikum Schwerin, Schwerin
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Universitätsklinikum Würzburg, Würzburg
- Greece (10):
  - Laiko General Hospital of Athens, Ampelokipoi
  - Henry Dunant Hospital, Athens
  - Metropolitan Hospital - First Oncology Clinic, Athens
  - Metropolitan Hospital - Fourth Oncology Clinic, Athens
  - Pepagni Hospital, Heraklion
  - Medical Center of Athens, Marousi
  - Interbalkan Medical Center of Thessaloniki, Pylaia
  - Theageneio Anticancer Oncology Hospital of Thessaloniki, Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
  - Bioclinic Thessaloniki (Galinos clinic), Thessaloniki
- Israel (6):
  - HaEmek Medical Center, Afula
  - Soroka University Medical Centre, Beersheba
  - Rambam Medical Center - PPDS, Haifa
  - Hadassah Medical Center - PPDS, Jerusalem
  - Rabin Medical Center - PPDS, Petah Tikva
  - Sheba Medical Center - PPDS, Ramat Gan
- Italy (11):
  - IRCCS Giovanni Paolo II Istituto Oncologico, Bari
  - ASST Papa Giovanni XXIII - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Fondazione del Piemonte per l'Oncologia (IRCCS), Candiolo
  - Ospedale Policlinico San Martino, Genova
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori IRST - PPDS, Meldola
  - Istituto Europeo Di Oncologia, Milan
  - Istituto Nazionale Dei Tumori, Milan
  - Azienda Ospedaliero Universitaria Di Modena Policlinico, Modena
  - Istituto Nazionale Per Lo Studio E La Cura Dei Tumori Fondazione Giovanni Pascale, Napoli
  - Istituto Oncologico Veneto - I.R.C.C.S., Padua
  - Azienda Ospedaliera Universitaria Senese, Siena
- Netherlands (8):
  - VU Medisch Centrum, Amsterdam
  - Zuyderland Medisch Centrum, Heerlen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Maxima Medisch Centrum, Veldhoven
  - Isala Klinieken, Zwolle
- New Zealand (5):
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Auckland City Hospital, Heidelberg
  - Tauranga Hospital, Tauranga
  - Wellington Hospital, Wellington
- Poland (5):
  - Bialostockie Centrum Onkologii im. Marii Sklodowskiej-Curie w Bialymstoku, Bialystok
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - NZOZ NEUROMED M. I M. Nastaj Spolka Partnerska, Lublin
  - Szpital Kliniczny im. Heliodora Swiecickiego w Poznaniu, Poznan
- Portugal (5):
  - Centro Hospitalar E Universitário de Coimbra EPE, Coimbra
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, E.P.E., Lisbon
  - Centro Hospitalar Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Hospital CUF Tejo, Lisbon
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe - PPDS, Porto
- Romania (4):
  - Affidea Romania SRL, Bucharest
  - S.C. Medisprof SRL, Cluj-Napoca
  - S.C. Onco Clinic Consult SA, Craiova
  - Oncology Center Sfantul Nectarie, Craiova
- Russia (9):
  - Chelyabinsk Regional Clinical Oncology Dispensary, Chelyabinsk
  - Clinical Oncology Centre #1, Krasnodar
  - Krasnoyarsk Regional Oncology Center n.a. A.I. Kryzhanovskiy, Krasnoyarsk
  - Kursk Regional Oncology Centre, Kursk
  - PMI Euromedservice, Pushkin
  - Ryazan Regional Clinical Oncology Dispensary, Ryazan
  - FSBI National Medical Research Center of Oncology n.a. N.N.Petrov of MHRF, Saint Petersburg
  - Railway Clinical Hospital JSC RZhD, Saint Petersburg
  - Regional Clinical Oncology Hospital, Yaroslavl
- Spain (15):
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Dexeus - Grupo Quironsalud, Barcelona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Córdoba
  - Hospital Universitario Virgen de La Arrixaca, El Palmar
  - Hospital Universitario de Jaen, Jaén
  - C.H. Regional Reina Sofia - PPDS, L'Hospitalet de Llobregat
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro - CIOCC, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Consorcio Hospital General Universitario de Valencia, Valencia
- United Kingdom (5):
  - Addenbrooke's Hospital, Cambridge
  - Castle Hill Hospital, Cottingham
  - Leicester Royal Infirmary, Leicester
  - Nottingham City Hospital, Nottingham
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eggermont AM, Ascierto PA, Khushalani NI, Schadendorf D, Boland G, Weber J, Lewis KD, Johnson D, Rivalland G, Khattak A, Majem M, Gogas H, Long GV, Currie SL, Chien D, Tagliaferri MA, Carlino MS, Diab A. PIVOT-12: a phase III study of adjuvant bempegaldesleukin plus nivolumab in resected stage III/IV melanoma at high risk for recurrence. Future Oncol. 2022 Mar;18(8):903-913. doi: 10.2217/fon-2021-1286. Epub 2022 Jan 25. PMID 35073733

RESULTS

PARTICIPANT FLOW:
Groups:
- Bempegaldesleukin (NKTR-214) + Nivolumab: Arm A: bempegaldesleukin (NKTR-214) 0.006 mg/kg intravenous (IV) infusion in combination with nivolumab 360 mg IV infusion (or 4.5 mg/kg IV infusion q3w for patients <40 kg) were administrated every 3 weeks q3w).
- Nivolumab: Arm B: Nivolumab 480 mg IV infusion (or 6.0 mg/kg IV infusion q4w for patients < 40 kg) every 4 weeks (q4w).
Period: Overall Study
Arm/Group | Bempegaldesleukin (NKTR-214) + Nivolumab | Nivolumab
Started | 378 | 387
Completed | 348 | 363
Not Completed | 30 | 24
Not completed — Lost to Follow-up | 3 | 9
Not completed — Withdrawal by Subject | 27 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bempegaldesleukin (NKTR-214) + Nivolumab | Nivolumab | Total
Number analyzed (Participants) | 378 | 387 | 765
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (14.21) | 56 (13.45) | 55.5 (13.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 148 | 310
  Male | 216 | 239 | 455
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 21 | 32
  Not Hispanic or Latino | 326 | 323 | 649
  Unknown or Not Reported | 41 | 43 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 354 | 357 | 711
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 22 | 27 | 49
Region of Enrollment [Number; unit: participants]
  Romania | 2 | 1 | 3
  United States | 66 | 75 | 141
  Czechia | 10 | 10 | 20
  United Kingdom | 5 | 8 | 13
  Portugal | 7 | 6 | 13
  Russia | 25 | 25 | 50
  Spain | 37 | 47 | 84
  Greece | 18 | 25 | 43
  New Zealand | 15 | 18 | 33
  Austria | 9 | 12 | 21
  Netherlands | 10 | 10 | 20
  Poland | 11 | 11 | 22
  Italy | 35 | 39 | 74
  Israel | 9 | 3 | 12
  Australia | 39 | 38 | 77
  France | 25 | 24 | 49
  Germany | 55 | 35 | 90
ECOG [Count of Participants; unit: Participants] — Measure Description: Eastern Cooperative Oncology Group (ECOG) performance status:
  ECOG Performance Status of 0 = Able to carry out all normal activities without restriction ECOG Performance Status of 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature
  Participants
    ECOG 0 | 351 | 351 | 702
    ECOG 1 | 27 | 36 | 63

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival (RFS) by Blinded Independent Central Review (BICR) of Bempegaldesleukin Plus Nivolumab Versus Nivolumab Alone.
Description: Recurrence-free Survival (RFS) of bempegaldesleukin plus nivolumab versus nivolumab alone is determined based on the disease recurrence date provided by Blinded Independent Central Review (BICR) and is defined as the time between date of randomization and date of first recurrence (local, regional, or distant metastasis by BICR), new primary melanoma (by BICR), or all-cause death, whichever occurs first.
Time Frame: Up to 21 months
Population: The study was terminated early due to the closure of the bempegaldesleukin clinical development program due to lack of enhanced efficacy being observed in combination with nivolumab therapy over nivolumab monotherapy for metastatic melanoma. As a consequence, no aggregate blinded independent central review data were collected; no comparative analyses between bempegaldesleukin + nivolumab arm vs nivolumab arm were conducted for this efficacy endpoint.
Arm/Group | Bempegaldesleukin (NKTR-214) + Nivolumab | Nivolumab
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Survival (OS) of Bempegaldesleukin Plus Nivolumab Versus Nivolumab Alone
Description: Overall Survival (OS) is defined as the time between the date of randomization and the date of death due to any cause. Patients who do not have a date of death will be censored on the last date for which a patient was known to be alive.
Time Frame: Up to 21 months
Population: For this outcome measure, the results were not estimable due to insufficient number of events. The study was terminated early due to the closure of the bempegaldesleukin clinical program due to lack of enhanced efficacy being observed in combination with nivolumab therapy over nivolumab monotherapy for metastatic melanoma. As a consequence, no comparative analyses between bempegaldesleukin + nivolumab arm vs nivolumab arm were conducted for this efficacy endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bempegaldesleukin (NKTR-214) + Nivolumab | Nivolumab
Number analyzed (Participants) | 378 | 387
months | NA [16.9 to NA] — Median and upper CI was not estimable due to insufficient number of events. | NA [NA to NA] — Median and 95% CI was not estimable due to insufficient number of events.

3. Secondary Outcome: Distant Metastasis-Free Survival (DMFS) by Investigator in Patients Who Are Stage III at Study Entry.
Description: Distant metastasis-free survival (DMFS) by Investigator is defined as the time between the date of randomization and the date of first distant metastasis by Investigator or date of death due to any cause, in patients who have Stage III melanoma at study entry.
Time Frame: Up to 21 months
Population: Participants include only patients who have Stage III melanoma at study entry. The results were not estimable due to insufficient number of events. The study was terminated early due to the closure of the bempegaldesleukin clinical development program due to lack of enhanced efficacy being observed in combination with nivolumab therapy over nivolumab monotherapy for metastatic melanoma.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bempegaldesleukin (NKTR-214) + Nivolumab | Nivolumab
Number analyzed (Participants) | 347 | 355
months | NA [NA to NA] — Median and 95% CI was not estimable due to insufficient number of events. | NA [NA to NA] — Median and 95% CI was not estimable due to insufficient number of events.

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: To evaluate safety and tolerability of (NKTR-214) 0.006 mg/kg in combination with nivolumab 360 mg IV infusion (or 4.5 mg/kg IV infusion q3w for patients <40 kg) and nivolumab 480 mg IV infusion (or 6.0 mg/kg IV infusion q4w for patients < 40 kg). Treatment-emergent adverse event (TEAE) is defined as an AE that was not present prior to treatment with study drug but appeared following treatment or was present at treatment start date but worsened during treatment-emergent period. The treatment-emergent period is defined as the period from the date of the first dose of study drug up to 30 days after the date of the last dose of study drug or the day prior to the initiation of subsequent anticancer treatment, whichever occurs first.
Time Frame: Approximately up to 21 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bempegaldesleukin (NKTR-214) + Nivolumab | Nivolumab
Number analyzed (Participants) | 378 | 387
Participants
  Patients who had a TEAE | 370 | 330
  Patients who had a Serious TEAE | 74 | 33
  Patients who had a TEAE of Grade 3 or higher | 120 | 50
  Patients who had a TEAE Leading to Death | 1 | 0

5. Secondary Outcome: Changes at 6 Months of Treatment From Baseline in Scores for the Global Health/Quality of Life (GH/QoL) and Physical Functioning Subscales of the European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire
Description: The EORTC QLQ-C30 comprises 30 items (i.e. single questions). 24 of which are aggregated into nine multi-item scales, that is, five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. Participants rate items and a score ranging from 0 to 100 is calculated. A higher score on the global health status/quality of life scale indicates a better level of functioning, and positive changes from baseline indicate improvement. A change of 5 - 10 points is considered a small change, and a change of 10 - 20 points is considered a moderate change. Due to the study termination, results for the mean change from baseline for GH/QoL and the physical functioning subscale were analyzed at approximately 6 months of treatment.
Time Frame: From baseline, up to approximately 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bempegaldesleukin (NKTR-214) + Nivolumab | Nivolumab
Number analyzed (Participants) | 378 | 387
score on a scale
  Global Health Status/QoL at Baseline | 79.20 (16.284) | 79.83 (15.698)
  Global Health Status/QoL at 6 Months | 77.31 (17.342) | 78.40 (16.776)
  Global Health Status/QoL Changes at 6 Months from Baseline | -3.71 (16.933) | -1.48 (16.921)
  Physical Functioning Subscale at Baseline | 91.81 (13.159) | 91.96 (13.515)
  Physical Functioning Subscale at 6 Months | 90.52 (12.417) | 91.16 (15.591)
  Physical Functioning Subscale Changes at 6 Months from Baseline | -2.41 (12.168) | -1.85 (13.861)

6. Secondary Outcome: Programmed Death-Ligand 1 (PD-L1) Expression as a Predictive Biomarker for Recurrence-free Survival (RFS)
Description: The predictive strength of Programmed Death-Ligand 1 (PD-L1) expression as a biomarker will be measured by the endpoint RFS by BICR based on PD-L1 expression level.
Time Frame: Up to 21 months
Population: as for outcome 1
Arm/Group | Bempegaldesleukin (NKTR-214) + Nivolumab | Nivolumab
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Recurrence-free Survival (RFS) by Investigator of Bempegaldesleukin Plus Nivolumab Versus Nivolumab Alone.
Description: Recurrence-free Survival by Investigator is defined as the time between the date of randomization and the date of first recurrence (local, regional, or distant metastasis by Investigator), new primary melanoma (by Investigator), or all-cause death, whichever occurs first.
Time Frame: Up to 21 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bempegaldesleukin (NKTR-214) + Nivolumab | Nivolumab
Number analyzed (Participants) | 378 | 387
months | NA [NA to NA] — Median and 95% CI was not estimable due to insufficient number of events. | NA [14.3 to NA] — Median and upper CI was not estimable due to insufficient number of events.

8. Secondary Outcome: Time to Disease Progression After the Next Line of Treatment for Study Patients Following Discontinuation of Bempegaldesleukin Plus Nivolumab Versus Nivolumab
Description: Time to disease progression after the next line of treatment is defined as time from randomization to progression per Investigator after the start of next line of therapy or death, whichever occurs first. Patients who were alive and without progression after the next line of therapy can be censored at last known alive date.
Time Frame: Up to 21 months
Population: The study was terminated early due to the closure of the bempegaldesleukin clinical development program due to lack of enhanced efficacy being observed in combination with nivolumab therapy over nivolumab monotherapy for metastatic melanoma. As a consequence, no data were collected for this efficacy endpoint.
Arm/Group | Bempegaldesleukin (NKTR-214) + Nivolumab | Nivolumab
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Distant Metastasis-Free Survival (DMFS) by Blinded Independent Central Review (BICR) in Patients Who Are Stage III at Study Entry.
Description: Distant Metastasis-Free Survival (DMFS) by Blinded Independent Central Review (BICR) is defined as the time between the date of randomization and the date of first distant metastasis by BICR or date of death due to any cause, whichever occurs first, in patients who have Stage III melanoma at study entry.
Time Frame: Up to 21 months
Population: The study was terminated early due to the closure of the bempegaldesleukin clinical development program due to lack of enhanced efficacy being observed in combination with nivolumab therapy over nivolumab monotherapy for metastatic melanoma. As a consequence, no blinded independent central review data were collected; no comparative analyses between bempegaldesleukin + nivolumab arm vs nivolumab arm were conducted for this efficacy endpoint.
Arm/Group | Bempegaldesleukin (NKTR-214) + Nivolumab | Nivolumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs will be reported starting immediately after the patient has been administered the first dose of study drug(s) until 100 days after the last dose of all study drug(s), up to a maximum of approximately 21 months. All ongoing non-serious AEs will be followed until resolution, the patient is lost to follow-up, patient death, or until the last Safety Follow-Up Visit. If the AE has not completely resolved by the last Safety Follow-Up Visit, the final outcome of these ongoing AEs will be captured.
Arm/Group | Combination of Bempegaldesleukin (NKTR-214) + Nivolumab | Nivolumab
All-Cause Mortality (participants affected / at risk) | 9/378 | 4/387
Serious Adverse Events (participants affected / at risk) | 74/378 | 33/387
Other Adverse Events (participants affected / at risk) | 369/378 | 329/387
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination of Bempegaldesleukin (NKTR-214) + Nivolumab (N=378) | Nivolumab (N=387)
Atrial fibrillation (Cardiac disorders) | 4 | 1
Myocarditis (Cardiac disorders) | 3 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pleuropericarditis (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Autoimmune myocarditis (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Autoimmune neuropathy (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Lacunar stroke (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Corona virus infection (Infections and infestations) | 3 | 2
Cellulitis (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infected seroma (Infections and infestations) | 1 | 0
Myelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 6 | 1
Chills (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 3 | 0
Hypersensitivity (Immune system disorders) | 2 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Autoimmune myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 1
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Eosinophilia (Blood and lymphatic system disorders) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Capillary permeability increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 1
Troponin T increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 0 | 1
Poor venous access (Vascular disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 2 | 1
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Thyroiditis (Endocrine disorders) | 1 | 1
Primary adrenal insufficiency (Endocrine disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 3 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Autoimmune nephritis (Renal and urinary disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Blindness transient (Eye disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination of Bempegaldesleukin (NKTR-214) + Nivolumab (N=378) | Nivolumab (N=387)
Pyrexia (General disorders) | 160 | 22
Fatigue (General disorders) | 154 | 112
Influenza like illness (General disorders) | 114 | 11
Asthenia (General disorders) | 70 | 38
Chills (General disorders) | 55 | 7
Face oedema (General disorders) | 21 | 1
Oedema peripheral (General disorders) | 21 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 95 | 54
Rash (Skin and subcutaneous tissue disorders) | 75 | 34
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 55 | 21
Erythema (Skin and subcutaneous tissue disorders) | 46 | 4
Pruritus generalised (Skin and subcutaneous tissue disorders) | 37 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 31 | 9
Nausea (Gastrointestinal disorders) | 106 | 50
Diarrhoea (Gastrointestinal disorders) | 101 | 68
Vomiting (Gastrointestinal disorders) | 52 | 17
Abdominal pain upper (Gastrointestinal disorders) | 34 | 12
Dry mouth (Gastrointestinal disorders) | 33 | 15
Abdominal pain (Gastrointestinal disorders) | 24 | 18
Constipation (Gastrointestinal disorders) | 23 | 27
Arthralgia (Musculoskeletal and connective tissue disorders) | 83 | 49
Myalgia (Musculoskeletal and connective tissue disorders) | 67 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 33 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 15
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 19 | 7
Headache (Nervous system disorders) | 85 | 46
Dizziness (Nervous system disorders) | 37 | 18
Paraesthesia (Nervous system disorders) | 20 | 4
Corona virus infection (Infections and infestations) | 49 | 47
Cough (Respiratory, thoracic and mediastinal disorders) | 52 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 | 14
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 22 | 4
Hyperthyroidism (Endocrine disorders) | 80 | 35
Hypothyroidism (Endocrine disorders) | 65 | 39
Alanine aminotransferase increased (Investigations) | 37 | 24
Aspartate aminotransferase increased (Investigations) | 27 | 22
Decreased appetite (Metabolism and nutrition disorders) | 53 | 13
Hypotension (Vascular disorders) | 40 | 3
Eosinophilia (Blood and lymphatic system disorders) | 45 | 7
Infusion related reaction (Injury, poisoning and procedural complications) | 25 | 9
Insomnia (Psychiatric disorders) | 26 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT04410445/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT04410445/SAP_001.pdf